CLINICAL TRIAL: NCT04597671
Title: NVALT 28/ PRL01 Durvalumab and Low-dose Prophylactic Cranial Irradiation (PCI) Versus Durvalumab and Observation in Radically Treated Patients With Stage III Non-small Cell Lung Cancer: A Phase III Randomized Study
Brief Title: Durvalumab and Low-dose PCI vs Durvalumab and Observation in Radically Treated Patients With Stage III NSCLC (NVALT28)
Acronym: NVALT28
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Association NVALT Studies (Other)
Responsible Party: Sponsor
Organization: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NVALT28
Record Dates: First submitted 2020-09-24; First posted 2020-10-22 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: PCI; immunotherapy; NSCLC; QoL
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Durvalumab with low-dose PCI
  Interventions: Drug: Durvalumab; Radiation: low-dose PCI
- Arm B (Active Comparator): Durvalumab with observation
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is used as standard of care
  Other Names: Imfinzi
Radiation: low-dose PCI — PCI will be given concurrently with durvalumab. PCI will be given to a dose of 15 Gy in 10 fractions
  Other Names: Prophylactic Cranial Irradiation (PCI)
  Arms: Arm A

SUMMARY:
This trial studies the combination of low-dose PCI with or without durvalumab in patients with radically treated stage III NSCLC. The hypothesis is that the incidence of brain metastases will be reduced from 30% to 15 % with durvalumab and to a maximum of 5% with the addition of low-dose PCI. This strategy would make brain metastases in stage III NSCLC history and this would improve QoL.

DETAILED DESCRIPTION:
The brain is frequently a site of disease relapse in Non-Small Cell Lung Cancer (NSCLC) patients. For radically treated patients, stage III has the highest risk for brain metastases with a cumulative incidence of brain metastases after radical treatment of approximately 30% for which there is no cure at the moment, decreasing the long-term survival and Quality of Life. Strategies to reduce incidence of brain metastases are necessary.

Prophylactic Cranial Irradiation (PCI) has been shown to reduce the incidence of brain metastases in patients with NSCLC. However, PCI leads to a neurocognitive impairment in about 25% of patients without altering the QoL.

The addition of durvalumab after chemo-radiotherapy in stage III NSCLC could reduce the incidence of brain metastases. In pre-clinical models, immunotherapy potentiates the effects of radiotherapy by a factor two to five. This makes the combination of PCI and immunotherapy interesting to evaluate whether it can further decrease the percentage of brain metastases as well as preserve organ function as a lower radiation dose can probably be used when combined with an antiprogrammed death (ligand)1 (PD(L)-1).

The hypothesis of the NVALT28 trial is that the combination of PCI with durvalumab will decrease the incidence of brain metastases from 30% to 15 % with durvalumab and to a maximum of 5% with the addition of low-dose PCI. This strategy would make brain metastases in stage III NSCLC history and this would improve QoL.

ELIGIBILITY:
Inclusion criteria:

1. Patients must sign a study-specific informed consent
2. TNM8 stage IIIA, IIIB or IIIC non-small cell lung cancer before start of concurrent chemoradiotherapy (preferentially histology; cytology is allowed)
3. Whole body FDG-PET-scan and brain imaging (MRI or CT with iv contrast) before the start of chemoradiotherapy: No distant metastases.
4. Additional brain MRI (MRI mandatory) dated within 28 days before randomization: no brain metastases.
5. Eligible for durvalumab treatment according to registration label of durvalumab in the Netherlands. Durvalumab has to be given in standard of care. (durvalumab has to be started already before randomization and PCI (i.e. at least one administration of durvalumab has to be given before randomization).
6. Treatment completed with concurrent chemoradiation. The last day of chemoradiotherapy should be within 80 days of randomization and randomization should be after start of durvalumab. Any platinum doublet or daily cisplatin regimen that is standard of care in The Netherlands is allowed. No disease progression after chemoradiotherapy (evaluated with CT-thorax and upper abdomen during/after the last dose of chemoradiotherapy and comparison with CT before start of chemoradiotherapy). Consolidation chemotherapy cycles after radiotherapy is not permitted but administration of 1 cycle of chemotherapy prior to concurrent chemo-radiotherapy is acceptable. Where possible, chemotherapy regimens should be given according to National Comprehensive Cancer Network (NCCN) Guidelines or European Society for Medical Oncology (ESMO) Guidelines.
7. To be eligible for randomization, patients must have received a total dose of thoracic radiotherapy of 60-66 Gy in 2 - 2.75 Gy per day, oncedaily fractions, or in case of daily cisplatin regimen 60.5-66 Gy in 22-24 fractions. Other radiotherapy schedules are not allowed. Sites are encouraged to adhere to the organ at risk constraints as used in the PACIFIC study as well as the EORTC recommendations for high-dose radiotherapy for lung cancer:

   1. Mean lung dose must be <20 Gy and/or V20Gy must be <35%
   2. Mean oesophagus dose must be <34 Gy
   3. Heart V45Gy <35% or V30Gy <30%.
8. Proton therapy to the chest is allowed.
9. ECOG performance status 0-1 at the time of randomization.
10. Evidence of postmenopausal status, or negative urinary or serum pregnancy test for female premenopausal patients.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 4 weeks.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or a study that will not influence the primary and secondary endpoint parameters (e.g. bioimpedance measurements, E-Nose) or the follow-up period of an interventional study. Note: participation in the NVALT31 study (follow up with CT thorax or PET-CT) is allowed
3. Mixed small cell and non-small cell lung cancer histology.
4. Patients who receive sequential chemoradiation therapy for locally advanced NSCLC.
5. Disease progression after completion of definitive platinum based, concurrent chemoradiation therapy, as proven by a CT scan after end of chemoradiation.
6. Any unresolved toxicity CTCAE (v. 5.0) more than grade 2 (i.e. grade 3 or higher) from the prior chemoradiation therapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by PCI may be included (e.g. hearing loss) after consultation with the principal investigator.
7. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment.
8. Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, diabetes type I or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
9. Active or prior documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis).
10. History of primary immunodeficiency.
11. History of organ transplant that requires therapeutic immunosuppression.
12. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses or psychiatric illness/ social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent.
13. Known history of tuberculosis, hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV).
14. History of another primary malignancy within 2 years prior to starting study drug, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study.
15. Prior cranial irradiation is not allowed.
16. Except for durvalumab after concurrent chemoradiotherapy, no previous treatment with PD-(L)1-inhibitors is allowed.
17. Female patients who are pregnant, breastfeeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
18. Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of incidence of brain metastases | From randomisation until moment of discovery of brain metastases or latest at 24 months after randomization
  To evaluate whether the addition of PCI to durvalumab after concurrent chemo-radiotherapy for stage III NSCLC reduces the cumulative incidence of brain metastases.

SECONDARY OUTCOMES:
Effect on neurocognitive functioning | From randomization until 24 months after randomization
  To evaluate what the effect is on neurocognitive functioning to be meassured with HVLT-R carried out by hospital staff.
Time to develop neurological symptoms | From randomization until time to develop neurological symptoms with a maximum of 24 months after randomization
  To evaluate time to develop neurological symptoms (CTCAE version 5.0)
Toxicity assessment | From randomization until end of study treatment
  To evaluate adverse events (CTCAE v 5.0 and PRO-CTCAE) that is the result of study treatment
Patient reported neurocognitive decline | From randomization until 5 years after randomization
  To evaluate patient reported neurocognitive decline using PRO-CTCAE (patient reported outcome)
Cost-efficiency | From randomization until end of study treatment
  To evaluate cost-efficiency of the addition of PCI to durvalumab with a state-transition model, calculated with Dutch tariff

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD PhD, Principal Investigator — Maastricht University/ Maastro clinic; Lizza Hendriks, MD PhD, Principal Investigator — Maastricht UMC
Locations (14):
- Netherlands (14):
  - ZGT, Almelo
  - AmsterdamUMC - location VUmc, Amsterdam
  - Radiotherapie Groep, Arnhem
  - Rijnstate, Arnhem
  - Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - ZRTI, Flushing
  - UMCG, Groningen
  - Maastro, Maastricht
  - Canisius Wilhemina Ziekenhuis, Nijmegen
  - Radboud UMC, Nijmegen
  - ZorgSaam Ziekenhuis, Terneuzen
  - Maxima Medisch Centrum, Veldhoven
  - Zaans Medisch Centrum, Zaandam

IPD SHARING:
Plan to Share IPD: No